CLINICAL TRIAL: NCT02152072
Title: Using Simulation-Based Training to Incorporate Lung Ultrasound Into Physical Examination
Status: Withdrawn | Type: Observational
Why Stopped: No Participant Enrolled
Sponsor: Tulane University Health Sciences Center (Other)
Responsible Party: Principal Investigator, Fayez Kheir,MD,MSc, Assistant Professor of Medicine,Department of Pulmonary and Critical Care, Tulane University Health Sciences Center
Organization: Tulane University (Other)
Other Study IDs: 609459-1
Record Dates: First submitted 2014-05-22; First posted 2014-06-02 (Estimated); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Medical Students,Lung Ultrasound,Simulation Training

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- medical students
  Interventions: Other: Using Simulation-Based Training to Incorporate Lung Ultrasound into Physical Examination

INTERVENTIONS:
Other: Using Simulation-Based Training to Incorporate Lung Ultrasound into Physical Examination

SUMMARY:
Dyspnea is a common symptom encountered frequently by medical practitioners. The differential diagnosis for a patient with such a symptom is broad and time consuming, while immediate management for distressed patients is what is desired. Lung ultrasound (LUS) is a relatively new technique that will help physicians more accurately diagnose and manage patients who present with dyspnea.

Focused medical ultrasonography education is becoming integrated into many physician residency training programs. Recent studies indicate a possible relationship between focused ultrasonography training in medical school curricula and improved physical examination accuracy. Thus, a short-term training program in LUS during medical school will have a major impact on physicians to be comfortable in using this skill when dealing with distressed patients in their prospective residency training. It will reduce educational burdens for physician residency programs and improve overall physician competency.

Simulation-based medical education (SBME) is ideally suited for offering effective training in a zero-risk environment. It enables trainees to gain knowledge and confidence in dealing with stressful clinical scenarios without exposing patients to any additional risk. SBME has also been shown to be a reliable tool for assessing learners' procedural skills and for teaching topics such as teamwork and communication.

The investigators hypothesize that simulation-based training of medical students will enable them to more effectively evaluate patients with shortness of breath using LUS.

ELIGIBILITY:
Inclusion Criteria:

* Third year medical students who signed the consent

Exclusion Criteria:

* a medical student who is not a third year and/or didn't signed the consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Medical Students
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Assess the pre and post-performance of medical students in using lung ultrasound (LUS) for patients with shortness of breath. | 8 weeks
  We designed the Thoracic Ultrasound Knowledge and Skills-Assessment Test (TUKSAT) which consists of questions about correctly identifying different organs using ultrasound (US) as well image acquisition skills as an objective measurement for students.
  Study participants will receive simulation-based LUS training through a course provided by a physician experienced in LUS as two sessions at the first week of their medical clerkship. TUKSAT as a pre-evaluation measure will be given.
  During the next 7 weeks, participants will be asked to see videos of LUS images where they will be asked to interpret the findings. A post-evaluation TUKSAT will then be given.

SECONDARY OUTCOMES:
Measure diagnostic agreement between trainees and experienced physicians in LUS following simulation-based medical education.. | 8 weeks
  Following their simulation-based training, participants will have videos of LUS images where they will be asked to interpret the findings. Diagnostic agreement will be compared between trainees' LUS finding and experienced physicians.

CONTACTS AND LOCATIONS:
Overall Officials: Fayez Kheir, MD,MSc, Principal Investigator — Tulane University